CLINICAL TRIAL: NCT01485393
Title: Pilot Study Comparing the Use of Dexmedetomidine and Zolpidem to Induce Natural Sleep
Brief Title: Polysomnographic Study Comparing the Use of Dexmedetomidine and Zolpidem to Induce Natural Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Assistant in Anesthaesia, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011P-000715; DP1OD003646 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Zolpidem

STUDY DESIGN:
Intervention Model Description: Patients will receive both interventions in a randomized order.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Control Subjects: Zolpidem, Then Dexmedetomidine (Experimental): This arm will enroll healthy control subjects, who will receive a regular nights sleep followed by a night of Zolpidem induced-sleep and then a night of Dexmedetomidine induced-sleep.
  Interventions: Drug: Dexmedetomidine; Drug: Zolpidem
- Healthy Control Subjects: Dexmedetomidine, Then Zolpidem (Experimental): This arm will enroll healthy control subjects, who will receive a regular nights sleep followed by a night of Dexmedetomidine induced-sleep and then a night of Zolpidem induced-sleep.
  Interventions: Drug: Dexmedetomidine; Drug: Zolpidem

INTERVENTIONS:
Drug: Dexmedetomidine — A dose of dexmedetomidine will be administered at 1mcg/kg over 10 minutes. Subjects will never receive active drugs (Zolpidem or dexmedetomidine concurrently).
  Other Names: Precedex
Drug: Zolpidem — 12.5 mg of oral Ambien CR. Subjects will never receive active drugs (Zolpidem/Ambien or dexmedetomidine concurrently).

SUMMARY:
The purpose of this study is to determine whether dexmedetomidine can be used to induce normal physiological sleep in humans.

ELIGIBILITY:
Inclusion Criteria:

* Primary Inclusion Criteria for "Insomniac" subjects:

Subjects will be deemed "Insomniacs" if they suffer from any of the following:

1. Subject will be required to meet the criteria for insomnia, set by the International Classification of Sleep Disorders, which requires that a patient have difficulty initiating or maintaining sleep that is not accounted for by another sleep disorder, neurologic or psychiatric disorder or substance or medication.
2. Subject will be required to not be on any current pharmacological sleep disorder treatment.
3. Between the ages of 18 and 35 years.
4. Not taking any prescription medications that alter sleep, cognitive functions, or both.

Exclusion Criteria:

Primary Exclusion Criteria for "Healthy" control subjects:

1. Abnormal sleep habits:

   * sleeping less than 5 hours each night;
   * going to sleep before 9:00 PM or after 2:00 AM on a regular basis; or
   * Waking up before 5:00 AM or after 10:00 AM on a regular basis. This will be objectively assessed by wrist actigraphy measured for a 1-week duration prior to the first study night.
2. A sleep latency greater than 60 minutes, greater than 3 awakenings per night. This will also be objectively assessed by wrist actigraphy.
3. A score greater than or equal to 10 on the Epworth Sleepiness Scale.
4. Takes medication that alters sleep, cognitive function, or both.
5. Has a history of a known neurological or psychiatric problem.
6. Younger than 18 or older than 35 years of age.
7. Known or suspected sleep disorder(s).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Control Subjects: Zolpidem, Then Dexmedetomidine | Healthy Control Subjects: Dexmedetomidine, Then Zolpidem
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants who were either randomized to receive either Dexmedetomidine or Zolpidem initially.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 23.9 [21 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep Quality
Description: Sleep quality will be assessed objectively through EEG measures (changes from baseline in length of non-REM sleep, length of REM sleep, and length of N3 sleep--all assessed in minutes) and subjectively, utilizing a post sleep questionnaire to assess the difference in quantity of sleep (minutes) from baseline. Sleep quality is directly related to these measures of sleep quantity.
Time Frame: Approximately 8 hours
Population: All patients undergo both zolpidem- and dexmedetomidine-induced sleep. Data analysis for this cohort was performed irrespective of randomization order.
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Zolpidem-Induced Sleep: All healthy control subjects undergo a night of zolpidem-induced sleep.
- Dexmedetomidine-Induced Sleep: All healthy control subjects undergo a night of dexmedetomidine-induced sleep.
Arm/Group | Zolpidem-Induced Sleep | Dexmedetomidine-Induced Sleep
Number analyzed (Participants) | 10 | 10
minutes
  Changes in total non-REM sleep | 33.2 [4.6 to 61.7] | 0 [0 to 0]
  Changes in REM sleep | -35 [-60.3 to -9.8] | 0 [0 to 0]
  Changes in N3 sleep | 35.8 [2.7 to 68.9] | 26.8 [2.2 to 51.3]
  Subjective differences in sleep | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: Performance on a Psychomotor Vigilance Test (PVT) After Waking up From Sleep
Description: The PVT is a measure of reaction time. It is measured as Lapse 400, which is the number of responses on the PVT greater than 400 milliseconds.
Time Frame: Approximately 30 minutes after waking up
Population: as for outcome 1
Measure: Number; unit: responses
Arm/Group | Zolpidem-Induced Sleep | Dexmedetomidine-Induced Sleep
Number analyzed (Participants) | 10 | 10
responses | 26 | 12

ADVERSE EVENTS:
Time Frame: Through completion of all three study visits (approximately 2 weeks).
Groups:
- Zolpidem: This arm reflects the night of Zolpidem-induced sleep for all 10 participants.
- Dexmedetomidine: This arm reflects the night of Dexmedetomidine-induced sleep for all 10 participants.
Arm/Group | Zolpidem | Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Insomniac patients were not conducted as originally proposed due to difficult enrollment.

The Motor Sequence Task was not performed as originally proposed, so it has been removed as a secondary outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT01485393/Prot_SAP_000.pdf